CLINICAL TRIAL: NCT06558370
Title: Bladder Filling for Pain Relief in Nullliparous Patients Undergoing Diagnostic Office Hysteroscopy
Brief Title: Bladder Distension for Pain Relief in Nullliparous Patients Undergoing Diagnostic Office Hysteroscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Bedaya Hospital (Other)
Responsible Party: Principal Investigator, Usama M Fouda, Prof., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hysteroscopy/full bladder
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Hysteroscopy
Keywords: Hysteroscopy; Full bladder; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empty bladder group (Active Comparator): Patients in the empty bladder group will be instructed to empty the bladder immediately before the procedure. A colleague will perform transabdominal ultrasound to confirm that the bladder is empty.
  All the procedures will be performed using the vaginoscopic technique. A rigid 2.9-mm hysteroscope with a 30° lens and a 5-mm outer sheath (Karl Storz GmbH, Tuttlingen, Germany) will be used in all procedures.
  Interventions: Other: Empty bladder group
- Bladder distension group (Active Comparator): Patients in the bladder distension group will be instructed to drink one liter of water and to avoid urination during a period of 2 h before the scheduled procedure. A colleague will perform transabdominal ultrasound to confirm that the bladder is distended .
  All the procedures will be performed using the vaginoscopic technique. A rigid 2.9-mm hysteroscope with a 30° lens and a 5-mm outer sheath (Karl Storz GmbH, Tuttlingen, Germany) will be used in all procedures.
  Interventions: Other: Bladder distension group

INTERVENTIONS:
Other: Empty bladder group — Patients in the empty bladder group will be instructed to empty the bladder immediately before the procedure. A colleague will perform transabdominal ultrasound to confirm that the bladder is empty.
  All the procedures will be performed using the vaginoscopic technique. A rigid 2.9-mm hysteroscope with a 30° lens and a 5-mm outer sheath (Karl Storz GmbH, Tuttlingen, Germany) will be used in all procedures.
  Arms: Empty bladder group
Other: Bladder distension group — Patients in the bladder distension group will be instructed to drink one liter of water and to avoid urination during a period of 2 h before the scheduled procedure. A colleague will perform transabdominal ultrasound to confirm that the bladder is distended .
  All the procedures will be performed using the vaginoscopic technique. A rigid 2.9-mm hysteroscope with a 30° lens and a 5-mm outer sheath (Karl Storz GmbH, Tuttlingen, Germany) will be used in all procedures.
  Arms: Bladder distension group

SUMMARY:
This study is conducted to assess whether the passive uterine straightening of the uterus by means of bladder filling is associated with less pain experienced by nulliparous women during office hysteroscopy.

DETAILED DESCRIPTION:
A randomized controlled study revealed that bladder filling before office hysteroscopy was associated with less pain experienced by parous women . On the other hand, a randomized study revealed that misoprostol was more effective than bladder filling in minimizing the pain experienced by postmenopausal women during office hysteroscopy. Till now , no studies were conducted to detect the effect of bladder filling on the pain experienced by nulliparous women during office hysteroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparity

Exclusion Criteria:

* Parous patients
* Cervical pathology
* Previous cervical surgery
* Severe vaginal bleeding.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Intensity of pain | Immediately after the procedure
  Measured using 100 mm visual analogue scale ( 0 = no pain and 100 = worst possible pain)

CONTACTS AND LOCATIONS:
Overall Officials: Usama M Fouda, Prof., Principal Investigator — Cairo University
Locations (1):
- Obstetrics &Gynecology Department , Faculty of medicine ,Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fouda UM, Elshaer HS, Elsetohy KA, Youssef MA. Misoprostol versus uterine straightening by bladder distension for pain relief in postmenopausal patients undergoing diagnostic office hysteroscopy: a randomised controlled non-inferiority trial. Eur J Obstet Gynecol Reprod Biol. 2016 Aug;203:326-30. doi: 10.1016/j.ejogrb.2016.06.024. Epub 2016 Jul 1. PMID 27481125